CLINICAL TRIAL: NCT01993875
Title: A Randomized, Placebo-controlled, Double-blinded, Multicenter Study of the Pharmacodynamics, Pharmacokinetics, and Tolerability of a Liquid Form of Lubiprostone in Adult Subjects With Chronic Idiopathic Constipation
Brief Title: Pharmacodynamic, Pharmacokinetic, and Tolerability Study of a Liquid Form of Lubiprostone in Adult Subjects With Chronic Idiopathic Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Collaborators: Sucampo Pharma Americas, LLC (Industry); Takeda (Industry); Sucampo AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCMP-0211-301
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2015-07

CONDITIONS: Chronic Idiopathic Constipation
MeSH Terms: interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lubiprostone (Experimental)
  Interventions: Drug: Lubiprostone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lubiprostone — Liquid formulation, 12 mcg x 2 pumps administered orally twice daily (BID)
  Arms: Lubiprostone
Drug: Placebo — Matching liquid placebo, 0 mcg x 2 pumps administered orally twice daily (BID)
  Arms: Placebo

SUMMARY:
To evaluate the pharmacodynamics and tolerability of a liquid formulation of lubiprostone, as compared to matching placebo, when administered orally to subjects with chronic idiopathic constipation. Additionally, liquid formulation pharmacokinetics, including a comparison of fed and fasted pharmacokinetics, of the liquid formulation will be performed in a subset of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Medically-confirmed diagnosis of chronic idiopathic constipation
* Willing to discontinue use of prescribed or over-the-counter (OTC) medication that affects gastrointestinal motility during the study
* Stable dose of selective serotonin re-uptake inhibitors (SSRIs), serotonin-specific reuptake inhibitor (SNRIs), or monoamine oxidase inhibitors (MAO) inhibitors

Exclusion Criteria:

* Any gastrointestinal (GI) condition, other than constipation, affecting GI motility or defecation.
* Medical/surgical condition that might interfere with the absorption, distribution, metabolism, or excretion of the study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt
Locations (11):
- United States (11):
  - Anniston, Alabama
  - Anaheim, California
  - DeLand, Florida
  - Hollywood, Florida
  - Orlando, Florida
  - South Miami, Florida
  - Overland Park, Kansas
  - Marlton, New Jersey
  - Raleigh, North Carolina
  - Salt Lake City, Utah
  - West Bend, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lubiprostone: Participants received liquid formulation of Lubiprostone drug, 12 microgram (mcg) x 2 pumps administered orally twice daily (BID).
- Placebo: Participants received placebo matching the liquid formulation of Lubiprostone drug via pump administered orally BID.
Period: Overall Study
Arm/Group | Lubiprostone | Placebo
Started | 82 | 82
Completed | 75 | 76
Not Completed | 7 | 6

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) Population included all participants who received at least 1 dose of study medication.
Groups:
- Lubiprostone: Participants received liquid formulation of Lubiprostone drug, 12 mcg x 2 pumps administered orally BID.
- Total: Total of all reporting groups
Arm/Group | Lubiprostone | Placebo | Total
Number analyzed (Participants) | 82 | 82 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 75 | 153
  >=65 years | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (12.51) | 45.0 (12.82) | 46.1 (12.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 58 | 113
  Male | 27 | 24 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29 | 29 | 58
  Not Hispanic or Latino | 53 | 53 | 106
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 38 | 80
  White | 38 | 40 | 78
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 82 | 82 | 164
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 29.5 (5.03) | 30.9 (6.50) | 30.2 (5.84)
Previous AMITIZA use at randomization [Count of Participants; unit: Participants]
  No | 80 | 81 | 161
  Yes | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Spontaneous Bowel Movements (SBMs) Within 1 Week
Description: SBM is defined as any bowel movement (BM) that did not occur within the 24-hour period following use of a rescue medication.
Time Frame: within 1 week
Population: Modified Intention to Treat (mITT), defined as all participants who received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: number of SBMs
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 82 | 82
number of SBMs | 4.6 (3.33) | 4.0 (3.50)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority; p = 0.1290, ANCOVA — Treatment p-value is from an analysis of co-variance (ANCOVA) using the SBM rate as the dependent variable, treatment as fixed effect, and baseline rate as random effect

2. Secondary Outcome: Consistency of SBMs at Week 1
Description: Stool consistency was rated according to the 7-point Bristol Stool Form Scale: Type 1 = separate hard lumps, like nuts (hard to pass), Type 2 = sausage-shaped but lumpy, Type 3 = like a sausage but with cracks on the surface, Type 4 = like a sausage or snake, smooth and soft, Type 5 = soft blobs with clear-cut edges (passed easily), Type 6 = fluffy pieces with ragged edges, a mushy stool, Type 7 = watery, no solid pieces; entirely liquid.
Time Frame: at Week 1
Population: mITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 82 | 82
score on a scale | 3.2 (3.12) | 2.4 (3.38)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority; p = 0.1290, ANCOVA — Treatment p-value is from an ANCOVA using the SBM rate as the dependent variable, treatment as fixed effect, and baseline rate as random effect

3. Secondary Outcome: Overall Stool Consistency at Week 1
Description: Overall stool consistency was rated according to the 7-point Bristol Stool Form Scale: Type 1 = separate hard lumps, like nuts (hard to pass), Type 2 = sausage-shaped but lumpy, Type 3 = like a sausage but with cracks on the surface, Type 4 = like a sausage or snake, smooth and soft, Type 5 = soft blobs with clear-cut edges (passed easily), Type 6 = fluffy pieces with ragged edges, a mushy stool, Type 7 = watery, no solid pieces; entirely liquid.
Time Frame: at Week 1
Population: mITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 82 | 82
score on a scale | 3.3 (1.38) | 3.0 (1.17)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority; p = 0.2177, ANCOVA — Treatment p-value is from an ANCOVA using the mean stool consistency score as the dependent variable, treatment as fixed effect, and the baseline consistency score as random effect

4. Secondary Outcome: Mean Change From Baseline in Stool Consistency at Week 1
Description: Stool consistency was rated according to the 7-point Bristol Stool Form Scale: Type 1 = separate hard lumps, like nuts (hard to pass), Type 2 = sausage-shaped but lumpy, Type 3 = like a sausage but with cracks on the surface, Type 4 = like a sausage or snake, smooth and soft, Type 5 = soft blobs with clear-cut edges (passed easily), Type 6 = fluffy pieces with ragged edges, a mushy stool, Type 7 = watery, no solid pieces; entirely liquid. The change from baseline was calculated as post-treatment value (mean) minus the baseline value (mean).
Time Frame: Baseline and Week 1
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 82 | 82
Units on a scale | 1.8 (0.91) | 1.9 (0.81)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority; p = 0.2177, ANCOVA — [p-value comment as in outcome 3, analysis 1]

5. Secondary Outcome: Overall Straining at Week 1
Description: Bowel straining was rated on a scale of 0 to 4 (0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe).
Time Frame: Week 1
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 82 | 82
Units on a scale | 1.8 (0.91) | 1.9 (0.81)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority; p = 0.0664, ANCOVA — Treatment p-value is from an ANCOVA using the mean straining score as the dependent variable, treatment as fixed effect, and the baseline straining score as random effect

6. Secondary Outcome: Mean Change From Baseline in Straining at Week 1
Description: Bowel straining was rated as 0 = absent, 1 = mild, 2 = moderate, 3 = severe, 4 = very severe. The change from baseline was calculated as post-treatment value minus the baseline value.
Time Frame: Week 1
Population: mITT Population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Lubiprostone | Placebo
Number analyzed (Participants) | 82 | 82
Units on a scale | -1.1 (0.94) | -0.8 (0.82)
Statistical Analysis 1: Comparison: Lubiprostone vs Placebo; Test type: Superiority; p = 0.0664, ANCOVA — Treatment p-value is from an ANCOVA using the mean straining score as the dependent variable, treatment as fixed effect, and the baseline mean score as random effect

ADVERSE EVENTS:
Time Frame: Up to 7 Weeks
Arm/Group | Lubiprostone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/82
Other Adverse Events (participants affected / at risk) | 21/82 | 15/82
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lubiprostone (N=82) | Placebo (N=82)
Nausea (Gastrointestinal disorders) | 9 | 1
Flatulence (Gastrointestinal disorders) | 7 | 6
Abdominal distension (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Headache (Nervous system disorders) | 6 | 9
Presyncope (Nervous system disorders) | 5 | 0
Dizziness (Nervous system disorders) | 2 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No